CLINICAL TRIAL: NCT06775002
Title: SERS-Based Serum Molecular Spectral Screening for Non-Small Cell Lung Cancer vs. Small Cell Lung Cancer: A Multicenter, Open-Label, Double-Blind, Independent Data Analysis Clinical Trial
Brief Title: SERS-Based Serum Molecular Spectral Screening for Lung Cancer Type
Status: Not yet recruiting | Type: Observational
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-042
Record Dates: First submitted 2025-01-07; First posted 2025-01-14 (Actual); Last update posted 2025-03-31 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer, Non-Small Cell; Lung Cancer Small Cell Lung Cancer (SCLC)
Keywords: SERS; Raman; NSCLC; SCLC; diagnostic model
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chest CT confirmed the presence of a pulmonary space-occupying lesion, which ultimately led to a lun: Chest CT confirmed the presence of a pulmonary space-occupying lesion, which ultimately led to a lung biopsy or surgical intervention. Pathology indicated a malignant lung tumor.
  Interventions: Diagnostic Test: Serum Raman spectroscopy intelligent diagnostic system

INTERVENTIONS:
Diagnostic Test: Serum Raman spectroscopy intelligent diagnostic system — 1. Screening interested participants should sign the appropriate informed consent (ICF) prior to completion any study procedures. 2. The investigator will review symptoms, risk factors, and other non-invasive inclusion and exclusion criteria. 3. The following is the general sequence of events during the 3 months evaluation period. 4. Completion of baseline procedures Participants were assessed for 3 months and completed all safety monitoring.

SUMMARY:
Lung cancer can be divided into two major categories: small cell lung cancer (SCLC) and non-small cell lung cancer (NSCLC), with NSCLC accounting for about 85% and SCLC about 15%. The prognoses of different types of lung cancer vary significantly. Early identification of different pathological types of lung cancer is crucial to the patient's prognosis.

Raman Spectrum (RS), as a non-invasive and highly specific molecular detection technique, can obtain information at the molecular level, thereby sensitively detecting changes in biomolecules related to tumor metabolism such as proteins, nucleic acids, lipids, and sugars. Surface-enhanced Raman spectroscopy (SERS), developed based on this technology, is one of the feasible methods for high-sensitivity biomolecular analysis.

In preliminary study, the investigators collected serum Raman spectral data from a cohort of 233 patients with malignant lung tumors and built a Raman intelligent diagnostic system for SCLC and NSCLC based on a machine learning model, achieving an accuracy rate of 80%. To obtain the highest level of clinical evidence and truly achieve clinical translation, this prospective, multicenter clinical study aims to validate the use of this intelligent diagnostic system for the early diagnosis of SCLC.

DETAILED DESCRIPTION:
1. Screening interested participants should sign the appropriate informed consent (ICF) prior to completion any study procedures.
2. The investigator will review symptoms, risk factors, and other non-invasive inclusion and exclusion criteria.
3. Completion of baseline procedures, participants were assessed for 30 days and completed all safety monitoring.
4. After completing the baseline assessment and confirming enrollment, participants will be given 2ml of fasting venous blood.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with Lung cancer meeting the criteria of TNM (Ninth Edition);
2. Participants are willing to participate in this study and follow the research plan;
3. Participants or legally authorized representatives can give written informed consent approved by the Ethics Review Committee that manages the website;.

Exclusion Criteria:

1. Participants with concomitant other malignant tumors;
2. Participants with missing baseline clinical data;
3. Participants with severe underlying pulmonary diseases (such as bronchiectasis, bronchial asthma, or COPD), or those with a history of occupational or environmental exposure to dust, mines, or asbestos;
4. Participants who are uncooperative or refuse to participate in the clinical trial later on.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chest CT confirmed the presence of a pulmonary space-occupying lesion, which ultimately led to a lung biopsy or surgical intervention. Pathology indicated a malignant lung tumor.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Estimated)
Dates: Start 2026-04-05 (Estimated); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
pathology | through study completion, an average of 1 year
  The final pathology results of the lung lesion biopsy or post-surgery
Diagnostic accuracy | through study completion, an average of 1 year
  Determine whether the enrolled lung cancer patients are small cell lung cancer or non-small cell lung cancer through the RAMAN intelligent diagnostic system

SECONDARY OUTCOMES:
Time to RAMAN diagnosis | up to 30 days
  The time to perform RAMAN testing and obtain diagnostic results after obtaining serum
Safety assessment Results | up to 30 days
  AEs and SAEs through Day 30